CLINICAL TRIAL: NCT05798637
Title: Role of Inflammation in the Pathogenesis of Frailty in the Elderly: Studies on the Contribution of Blood Platelets- PIPAF Platelets in the Pathogenesis of Ageing Associated Frailty
Brief Title: PIPAF Platelets in the Pathogenesis of Ageing Associated Frailty
Acronym: PIPAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Paolo Gresele, Clinical Professor, Azienda Ospedaliera di Perugia
Other Study IDs: 3546/19
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus, Type 2; Alzheimer Disease
Keywords: Coronary Artery Disease; Diabetes Mellitus, Type 2; Alzheimer Disease; Platelets
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Alzheimer Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: Elderly subjects diagnosed with coronary syndrome ascertained by coronary angiography
  Interventions: Other: Standard of care
- Group B: Frail elderly
  Interventions: Other: Standard of care
- Group C: Elderly subjects with type 2 diabetes mellitus
  Interventions: Other: Standard of care
- Group D: Elderly subjects with alzheimer's disease
  Interventions: Other: Standard of care
- Group E: Not frail elderly subjects
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — No treatment other than clinical standard therapy is provided. Each subjects will perform a blood draw at enrollment and after 24 months of follow-up. Subjects will also be given a frailty status assessment questionnaire (according to the criteria of Fried)

SUMMARY:
This is a prospective observational study aimed at testing the existence of an association between frailty, inflammatory status, and degree of platelet activation and reactivity in elderly subjects with type 2 diabetes or coronary artery disease or Alzheimer's disease.

DETAILED DESCRIPTION:
Frailty in the elderly is a syndrome that strongly affects quality of life and represents a major social and economic challenge. Frailty often, and more frequently, occurs in individuals with aging-related diseases including type 2 diabetes, cardiovascular disease, and Alzheimer's disease. All of these diseases are associated with a state of weak chronic inflammation. Studies in recent years have pointed out that platelets can directly contribute to inflammatory processes. Due to of this ability to act as proinflammatory cells and of their strong involvement in various metabolic, cardiovascular, and neurodegenerative disorders, platelets appear to have key roles in the physio-pathological mechanisms that predispose to frailty.

In the present study, it is planned to recruit 4 cohorts of elderly patients, each of 40 patients, divided by pathology ( frail elderly, diabetic elderly, elderly with stable atherosclerotic coronary artery disease, elderly with early-stage Alzheimer's disease) and a cohort of 40 healthy elderly subjects. All subjects will perform a blood draw at enrollment and after 24 months of follow up in order to evaluate: the state of platelet activation; the aggregating response of platelets to stimuli such as thrombin, Adenosine DiPhosphate (ADP), and collagen; the state of chronic inflammation and oxidative stress; the procoagulant profile of platelets; presence of platelet subpopulations characterized by RNA, microRNA and/or protein profiling. Each subject will also be given a questionnaire to assess frailty status (according to Fried's criteria) and urine samples will be collected to perform the assay of metabolites such as 11dh-TXB, 8-hydroxy-2-deoxyguanosine (8-OHdG) and 8-epiPGF2a (8-isoprostane).

ELIGIBILITY:
Inclusion Criteria:

* age > 65 years
* low-dose aspirin therapy (100 mg)
* belonging to each of the cohorts indicated

Exclusion Criteria:

* Lack of inclusion criteria and/or consent to the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study involves 5 cohorts of patients:
  * patients diagnosed with stable ischemic heart disease (CAD)
  * frail elderly patients
  * patients with type 2 diabetes (T2DM)
  * patients with Alzheimer's disease (AD)
  * not frail elderly subjects (control group).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Rate of platelet activation | 3 years
  Platelet activation will be assessed in vivo, on circulating platelets, by flowcytometry measurement of p-selectin, integrin αIIbβ3, and tissue factor expression, and in vitro, on isolated platelets, by studying the response to agonists (thrombin, ADP, collagen) with lumiaggregometry and ATP secretion

SECONDARY OUTCOMES:
Rate of systemic inflammation and oxidative stress | 3 years
  Quantification of oxidative stress and chronic inflammation will be done by measuring the levels of 8-hydroxy-2-deoxyguanosine (8-OHdG) and 8-epiPGF2a (8-isoprostane) on urine and the levels of high-sensitivity PCR, sCD40L, sRAGE, TAT and F1+2 in plasma by enzyme immunoassay method.
Procoagulant platelet activity | 3 years
  Platelet procoagulant activity will be measured by quantifying thrombin generation from lysed platelets using the Calibrated Automated Thrombogram Assay
Rate of proinflammatory platelet activity | 3 years
  Proinflammatory platelet capacity will be estimated by measuring the expression of matrix metalloproteinases MMP-2 and MMP-9.
Rate of platelet heterogeneity | 3 years
  Platelets with procoagulant and proinflammatory activity will be identified by flowcytometry, and their transcripts/micro RNAs will be analyzed in the different patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gresele, Prof, Principal Investigator — University Of Perugia
Locations (2):
- Italy (2):
  - IRCCS Centro Cardiologico Monzino, Milan, Milan
  - Univeristà di Pavia, Pavia